CLINICAL TRIAL: NCT00236054
Title: A 10-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Flexible-Dosage Study to Evaluate the Efficacy and Safety of Gabitril (up to 16 mg/Day) in the Treatment of Adults With Generalized Anxiety Disorder
Brief Title: A 10-Week Efficacy and Safety Study for of Gabitril in the Treatment of Adults With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C6671/3032/AX/US
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Tiagabine

INTERVENTIONS:
Drug: Gabitril

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of an investigational anti-anxiety medication relative to placebo in patients with generalized anxiety disorder (GAD)

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 to 64 years of age (inclusive) will be eligible to participate if they satisfy the DSM-IV-TR criteria for GAD, as well as meeting the required screening and baseline visit scores for a series of psychiatric evaluations (i.e., HAM-A, HADS, MADRS and CGI-S).

Exclusion Criteria:

* Have been previously unresponsive to two or more adequate courses of pharmacological treatment for GAD
* Have been diagnosed with any other psychiatric Axis I disorder (except GAD) as a principal diagnosis within the past six months
* Have been diagnosed with any eating disorder within the past six months
* Have any history of OCD, psychotic disorder, bipolar disorder or antisocial personality disorder
* Have any history of alcohol or substance abuse within the past 3 months
* Have any history of seizures, including febrile seizures
* Have any history of head trauma associated with loss of consciousness within the past 15 years

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440
Dates: Start 2004-10; Study Completion 2005-12

PRIMARY OUTCOMES:
Reduction of symptomatology associated with Generalized Anxiety Disorder as assessed by the change from baseline to endpoint in the total score of the HAM-A scale.

SECONDARY OUTCOMES:
Assessment of proportion of responders and
patients in remission according to HAM-A scores and CGI ratings by
visit, assessment of the safety and tolerability in patients with GAD

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Pacific Institute for Medical Research, Inc., Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - Affiliated Research Institute, San Diego, California
  - Health Quest Clinical Trials, San Diego, California
  - Pacific Clinical Research Medical Group, Upland, California
  - UF Behavioral Health Clinic, Jacksonville, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Atlanta Institute of Medicine & Research - Atlanta Clinic, Atlanta, Georgia
  - Cunningham Clinical Research, LLC, Edwardsville, Illinois
  - LSUHSC Anxiety and Mood Disorders Clinic, New Orleans, Louisiana
  - Summit Research Network, Farmington Hills, Michigan
  - Social Psychiatry Research Inst., Brooklyn, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - Medical and Behavioral Health Research, PC, New York, New York
  - Hartford Research Group Ltd., Cincinnati, Ohio
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - South East Health Consultants, LLC, Charleston, South Carolina
  - Northwest Clinical Research Center, Bellevue, Washington
  - Northbrooke Research, Brown Deer, Wisconsin